CLINICAL TRIAL: NCT01959828
Title: Examination of Safety and Effectiveness of IK-3001 (Nitric Oxide for Inhalation) in Japanese Subjects With Pulmonary Hypertension Associated With Cardiac Surgery - Multi-Center, Open-Label, Clinical Study
Brief Title: Confirmatory Study of IK-3001 in Japanese Subjects With Peri-/Post-op Pulmonary Hypertension Assoc. With Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IK-3001-CVS-301
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension, Pulmonary; Ventricular Dysfunction, Left
Keywords: pulmonary hypertension; cardiac surgery; Glenn surgery; fontan surgery; left ventricular assist device; LVAD
MeSH Terms: conditions — Hypertension, Pulmonary; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- inhaled nitric oxide (Experimental): Adults: IK-3001 at start dose 20 ppm; may be increased to 40 ppm at the investigator's or subinvestigator's discretion (up to ~ 24 hrs).
  Children: IK 3001 at start 10 dose ppm; may be increased to 20 ppm at the investigator's or subinvestigator's discretion (up to ~24 hrs).
  Treatment with IK-3001 will continue until it is clinically indicated to begin the weaning process from IK-3001.
  Interventions: Drug: IK-3001

INTERVENTIONS:
Drug: IK-3001
  Other Names: inhaled nitric oxide

SUMMARY:
Sixteen Japanese subjects (6 adults/10 children) with peri- and post-operative pulmonary hypertension associated with cardiac surgery will be evaluated at approx. 6 sites for safety and efficacy of IK-3001.

DETAILED DESCRIPTION:
This is a multi-center, open-label, clinical study of the safety and efficacy of IK-3001 in 16 subjects with peri- and post-operative pulmonary hypertension associated with cardiac surgery. Two primary sub-sets of this patient population will be evaluated in this study:

1. Adults with severe congestive heart failure having LVAD implant
2. Children requiring surgery for congenital heart disease with corresponding PH or having Glenn surgery or Fontan surgery for single-ventricle physiology. Children with severe pulmonary hypertension due to congenital heart disease who require inhaled nitric oxide (iNO) pre-operatively may also be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must meet one of the following criteria:

   1. Adults, aged 15 to 80 years, with severe congestive heart failure (CHF) and scheduled for left ventricular assist device (LVAD) placement; or
   2. Children, aged < 15 years, scheduled for surgery for congenital heart disease which may associate pulmonary hypertension (PH)(including children with severe PH due to congenital heart failure and with severe hypoxemia secondary to high pulmonary vascular resistance or either a history or a possibility of developing PH crisis, who are deemed by an investigator or subinvestigator to require IK-3001 pre-operatively); or
   3. Children, aged < 15 years, with congenital heart disease and scheduled for Glenn surgery; or
   4. Children, aged < 15 years, with congenital heart disease and scheduled for Fontan surgery.
2. For women of childbearing potential, a negative result for a pregnancy test documented prior to enrollment.
3. Subjects must give written informed consent. If the subject is a minor the subject's legally acceptable representative (parent or legal guardian) must give written informed consent.

Exclusion Criteria:

1. Lung hypoplasia or other pre-existing severe lung disease;
2. Planned bi-ventricular support;
3. Participation in another clinical trial of an investigational agent within 28 days from the day of informed consent for this study including subjects who are deemed to carry a residual effect of an investigational product lasting more than 28 days from a previous investigational study;
4. Subjects with PH secondary to organic obstructive lesions in pulmonary arteries;
5. Subjects not under mechanical ventilation;
6. Investigator or subinvestigator decision that the subject is unsuitable for this study.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in mean pulmonary artery pressure (mPAP) in Adult subjects (with LVAD) | Predose baseline to 24 hours (or final observation, if < 24 hours) (measured at 1 hour, 4 hours, and 24 hours after initiation of IK-3001 therapy
Change in partial pressure of oxygen in arterial blood/fraction of inspired oxygen (PaO2/FiO2) ratio in Adult subjects (with LVAD) | Predose baseline to 24 hours (or final observation, if < 24 hours) (measured at 1 hour, 4 hours, and 24 hours after initiation of IK-3001 therapy
Change in central venous pressure (CVP) in Children (with congenital heart disease) | Predose baseline to 24 hours (or final observation, if < 24 hours)(measured at 1 hour, 4 hours, and 24 hours after initiation of IK-3001 therapy
Change in partial pressure of oxygen in arterial blood/fraction of inspired oxygen (PaO2/FiO2) ratio in Children (with congenital heart disease) | Predose baseline to 24 hours (or final observation, if < 24 hours) (measured at 1 hour, 4 hours, and 24 hours after initiation of IK-3001 therapy

CONTACTS AND LOCATIONS:
Overall Officials: Khurram Jamil, MD, Study Director — Mallinckrodt
Locations (7):
- Japan (7):
  - Osaka University Hospital, Osaka
  - National Cerebral and Cardiovascular Center (Pediatric CV Surgery), Osaka
  - National Cerebral and Cardiovascular Center (Transplantation), Osaka
  - The University of Tokyo Hospital, Tokyo
  - National Center for Child Health and Development, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Tokyo